CLINICAL TRIAL: NCT04401774
Title: Phase II Maintenance Trial of Nivolumab for Newly Diagnosed PCNSL Patients With Persistent Circulating Tumor DNA in the CSF After Completion of Methotrexate-Based First-Line Induction Chemotherapy
Brief Title: Nivolumab Maintenance in Newly Diagnosed PCNSL With Persistent CSF Circulating Tumor DNA After Completion of First-Line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-383
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL)
Keywords: Nivolumab; Persistent Circulating Tumor DNA; Methotrexate-Based First-Line Induction Chemotherapy; 19-383
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: The phase II nivolumab maintenance trial is an open-label trial for patients who have completed high-dose methotrexate-based first-line chemotherapy for primary central nervous system lymphoma (PCNSL) but have persistent cfDNA in their CSF after treatment despite imaging response.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab Maintenance (Experimental): All patients will undergo cerebrospinal fluid (CSF) and blood collection as well as MRI imaging as standard of care prior to (- 21 days) first-line treatment initiation, during first-line therapy (before initiation of the 5th methotrexate dose (+/- 7 days)), at completion of first-line chemotherapy therapy (+/- 7 days) as well as 60, 180, and 360 days after enrollment into maintenance or observation (+/- 7 days). Those patients with persistent cfDNA in the CSF after completion of first-line chemotherapy and either complete or partial response on imaging will be enrolled into the nivolumab maintenance treatment arm. All other patients (no persistent cfDNA in the CSF and either complete or partial response on imaging) are followed with observation. Patients who do not respond to first-line therapy are not eligible for nivolumab maintenance and will no longer be followed in the biospecimen and clinical data collection cohort.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be given every 4 weeks at 480mg flat dose intravenously for one year (total of 13 nivolumab doses).

SUMMARY:
The purpose of this additional part of the study is to test whether the study drug, nivolumab, is a safe treatment that will prevent participants' primary central nervous system lymphoma (PCNSL) from growing again (recurrence). Participants will be people with PCNSL who continue to have cell free tumor DNA (cfDNA) in their CSF despite completion of their first treatment (first-line treatment).

ELIGIBILITY:
Inclusion Criteria:

Biospecimen and Data Collection:

* Histologically documented PCNSL with the ability to submit up to 20 unstained formalinfixed, paraffin embedded (FFPE) slides from the initial tissue diagnosis prior to study registration or histologically confirmed lymphomatous involvement of the CSF and/or eye/vitreous
* Patients must be able to tolerate MRI/CT scans with [18F FDG]
* Patients must be able to tolerate lumbar punctures and/or Ommaya taps

Additional Criteria for Nivolumab Maintenance Arm:

All criteria in the above "Biospecimen and Data Collection" section must be satisfied as well as:

* Persistent cfDNA in the CSF
* Participants must be able to understand and be willing to sign a written informed consent document
* Women and men who are at least 18 years of age on the day of consenting to the study
* KPS ≥60
* Life expectancy of > 3 months (in the opinion of the investigator)
* Participants must have adequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) ≥ 0.75 x 10^9/L
  * Platelets ≥ 75 x 10^9/L and no platelet transfusion within the past 21 days prior to study registration
  * Hemoglobin (Hgb) ≥ 8 g/dL and no red blood cell (RBC) transfusion within the past 21 days prior to study registration
  * International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal. Patients on anticoagulants should be managed according to MSK SOPs as outlined in: 'Therapeutic Anticoagulation Guidelines in Adults' regarding management of anticoagulants prior to each CSF collection. Please discuss any complicated patient with the PI for consideration.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal
  * Serum bilirubin ≤ 1.5 times the upper limit of normal; or total bilirubin ≤ 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome
  * Serum creatinine ≤ 2 times the upper limit of normal
* Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 5 months after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 7 months after the last dose
* Women of childbearing potential must have a negative plasma pregnancy test upon study entry. See section on Pregnancy and Reproduction

Exclusion Criteria:

Biospecimen and Data Collection:

* Patients with recurrent/refractory PCNSL. Patients with stable disease as their best response to first-line chemotherapy will also come off study.
* Patient with systemic, non-CNS lymphoma metastatic to the CNS
* Patient is known to have human immunodeficiency virus (HIV) infection
* Patient is known to have a history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests
* Patient's who are planned to undergo consolidation with autologous HSCT

Additional Criteria for Nivolumab Maintenance Arm:

None of the criteria in the above "Biospecimen and Data Collection" section can be present. The following criteria must also not be present:

* Patient has undergone prior allogenic stem cell transplant
* Patient's who are planned to undergo consolidation with autologous HSCT
* Any chemotherapy, external beam radiation therapy, or anticancer antibodies within 14 days of the first dose of study drug
* Patient is allergic to components of the study drug
* Patient is concurrently using other approved or investigational antineoplastic agents
* Previous or current treatment with an anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PDL2 agent
* Patient has an active concurrent malignancy requiring active therapy
* Patient is requiring escalating or chronic supraphysiologic doses of corticosteroids (> 8 mg dexamethasone daily) for control of disease at the time of registration
* Patient is using systemic immunosuppressant therapy including: cyclosporine A, tacrolimus, sirolimus, and other such medications, or chronic administration of > 5 mg/day of prednisone or the equivalent. Participants must be off immunosuppressant therapy for at least 28 days prior to the first dose of the study drug
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Known history of, or any evidence of active, non-infectious pneumonitis
* Patient has significant abnormalities on screening electrocardiogram (EKG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, uncontrolled congestive heart failure, uncontrolled hypertension, valvular disease, pericarditis, or myocardial infarction within 6 months of screening
* Peptic ulcer, abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within past 6 months
* Patient is known to have an uncontrolled active systemic infection
* Patient has a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject's safety or put the study outcomes at undue risk
* Women who are pregnant or nursing (lactating), where pregnancy is defined as a state of a female after conception until the termination of gestation, confirmed by a positive plasma hCG laboratory test of > 5 mIU/mL (See section on Pregnancy and Reproduction)
* The patient is unwell or unable to participate in all required study evaluations and procedures
* Participants who have received a live / attenuated vaccine within 30 days of first treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
Frequencies of toxicities | within 60 days of therapy
  Frequencies of toxicities will be summarized based on the Common Toxicity Criteria (CTCAE) version 5.0. Adverse events.
cfDNA conversion rate in CSF | 12 months
  Conversion rate is defined as the proportion of patients receiving maintenance nivolumab who have undetectable cfDNA at one-year from the start of nivolumab maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grommes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm